CLINICAL TRIAL: NCT03958032
Title: Effects of Sarcopenia on Early Postoperative Outcomes in Patients Undergoing Surgical Treatment for Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali GUNER, Associate Professor, Karadeniz Technical University
Other Study IDs: sarcopenia01
Record Dates: First submitted 2019-05-18; First posted 2019-05-21 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Gastric Cancer; Sarcopenia; Malnutrition; Cachexia; Complication
Keywords: sarcopenia; cancer; gastrointestinal
MeSH Terms: conditions — Stomach Neoplasms; Sarcopenia; Malnutrition; Cachexia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with gastric cancer: All consecutive patients undergoing surgery due to gastric cancer will be included in this study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention is planned for the participants for the treatment of gastric cancer. Treatment decision will be in line with clinical practice guidelines. Surgical team will be blind to the participant's sarcopenia status.

SUMMARY:
We aimed to establish the effects of sarcopenia on postoperative complications among patients undergoing surgical treatment for gastric cancer

DETAILED DESCRIPTION:
Among gastrointestinal disease, gastric cancer is a malignancy which is diagnosed predominantly in advanced stages, mostly accompanied with malnutrition when diagnosed, has aggressive behavior with poor oncological outcomes. The only option for curative treatment is surgical resection in this malignancy; however, the surgical procedure itself causes high morbidity and mortality rates. Therefore, physicians combine various treatment modalities and risk assessment to decrease complication and mortality rates.

Sarcopenia is a syndrome characterized by progressive and generalized loss of skeletal muscle mass and strength with a risk of adverse outcomes such as physical disability, poor quality of life, and death. For the diagnosis of sarcopenia, using the presence of both low muscle mass and decreased muscle function (strength or performance) is recommended. Previous studies showed that colorectal or pancreatic cancer accompanied with sarcopenia has adverse effects on not only for short term and also for long term outcomes. The majority of studies regarding gastric cancer was published from Eastern countries owing to their high incidence. There are few studies from western countries which are mostly retrospective and does not meet the diagnostic criteria of sarcopenia. In the western population, there is no high-quality evidence so far regarding the impact of sarcopenia on early outcomes of gastric cancer surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing gastric surgery for gastric cancer
2. Histologically proven gastric adenocarcinoma
3. Patients over 18 years
4. Patients who agreed to participate in the study

Exclusion Criteria:

1. patients treated by non-surgical treatment such as endoscopic treatment, palliative chemotherapy)
2. patients received palliative surgery without gastric resection (bypass procedures)
3. patients required thoracotomy/thoracoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing surgery due to gastric cancer will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2016-12-03 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | within 30 days after surgery
  complications graded by Clavien-Dindo Complication Classification System

SECONDARY OUTCOMES:
Length of hospital stay | up to 90 days
  time interval from the date of operation to the date of discharge
Mortality | within 30 days after surgery
  Dying after surgery
Readmission rate | within 30 days after surgery
  readmission to the hospital because of the adverse events after discharge
Incidence of sarcopenia | one day before surgery
  Sarcopenia consensus defined by The European Working Group on Sarcopenia in Older People
Muscle mass volume | one day before surgery
  muscle mass volume of a cross-sectional computerized- tomography image of the L3, corrected for patient height resulting in L3 muscle index.
Psoas muscle mass volume | one day before surgery
  muscle mass volume of Psoas muscle with 3D reconstruction
Muscle strength | one day before surgery
  evaluated by handgrip strength test (with digital dynamometer)
Physical performance | one day before surgery
  evaluated by 4-meter gait speed test
Major complication | within 30 days after surgery
  grade 3 or higher complications graded by Clavien-Dindo Complication Classification System

CONTACTS AND LOCATIONS:
Overall Officials: Ali GUNER, MD, Principal Investigator — Karadeniz Technical University Faculty of Medicine
Locations (1):
- Karadeniz Technical University, Faculty of Medicine, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Background] Fukuda Y, Yamamoto K, Hirao M, Nishikawa K, Nagatsuma Y, Nakayama T, Tanikawa S, Maeda S, Uemura M, Miyake M, Hama N, Miyamoto A, Ikeda M, Nakamori S, Sekimoto M, Fujitani K, Tsujinaka T. Sarcopenia is associated with severe postoperative complications in elderly gastric cancer patients undergoing gastrectomy. Gastric Cancer. 2016 Jul;19(3):986-93. doi: 10.1007/s10120-015-0546-4. Epub 2015 Sep 25. PMID 26407875
- [Background] Tegels JJ, van Vugt JL, Reisinger KW, Hulsewe KW, Hoofwijk AG, Derikx JP, Stoot JH. Sarcopenia is highly prevalent in patients undergoing surgery for gastric cancer but not associated with worse outcomes. J Surg Oncol. 2015 Sep;112(4):403-7. doi: 10.1002/jso.24015. Epub 2015 Aug 31. PMID 26331988
- [Background] Guner A. Recent trends of gastric cancer treatment in Turkey. Transl Gastroenterol Hepatol. 2017 Apr 26;2:31. doi: 10.21037/tgh.2017.04.01. eCollection 2017. PMID 28529985